CLINICAL TRIAL: NCT01985295
Title: Phase I Clinical Study of a Combined Modality Treatment of Sarcomas of the Extremities With Radiotherapy (RT) and Dose-escalation of Pazopanib
Brief Title: Combined Modality Treatment of Sarcomas of the Extremities
Acronym: PASART-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M09RTP; 2009-014901-15 (EudraCT Number)
Record Dates: First submitted 2013-10-07; First posted 2013-11-15 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cohort (Other): Dose level Dose of pazopanib orally, once daily, # patients -1 200 mg --
  1. (starting) 400 mg 3
  2. 600 mg 3
  3. (maximum) 800 mg 3
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — A dose escalation trial of Pazopanib, starting at 400mg daily, orally in combination with the standard 25 x 2Gy preoperative radiotherapy in newly diagnosed extremity sarcoma patients. Dose of pazopanib will be escalated via 600mg to maximally 800mg. Overall treatment time of pazopanib is 40 days.
  Other Names: Compound Number: GW786034

SUMMARY:
In this study, we aim to define the recommended dose of a VEGFR-TKI (pazopanib) in combination with RT pre-operatively given.

DETAILED DESCRIPTION:
Study design A dose escalation trial of Pazopanib, starting at 400mg daily, orally in combination with the standard 25 x 2Gy preoperative radiotherapy in newly diagnosed extremity sarcoma patients. Dose of pazopanib will be escalated via 600mg to maximally 800mg. Overall treatment time of pazopanib is 40 days.

Treatment plan: Pazopanib Dose level Dose of pazopanib orally, once daily, # patients

1. (starting) 400 mg 3
2. 600 mg 3
3. (maximum) 800 mg 3

Treatment plan: radiotherapy RT is given during 5 weeks with a once daily fraction of 2 Gray (50 Gray in 25 daily fractions)

RT planning: The dose planning should be performed by CT based Intensity Modulated RT (IMRT) or 3 Dimensional Conformal RT (3D-RT) according to the local planning protocol of the participating institute.

Dose specification: According to the ICRU 50/62.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed newly diagnosed intermediate to high grade soft tissue sarcoma of and localized to the extremities or head and neck area for which the treatment is a combination of both surgery and radiotherapy (deep seated, > 5cm according to the RECIST 1.1 criteria, grade II/III according to the WHO definition).
2. Age > 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
5. Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

6 Able to swallow and retain oral medication. 7. A life expectancy of at least 12 weeks. 8. Adequate organ function.

-

Exclusion Criteria:

1. Prior malignancies; except subjects who have had another malignancy and have been disease-free for 5 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
2. Patients with recurrent sarcomas (even without prior radiotherapy).
3. Ewing sarcoma and other PNET family tumours, rhabdomyosarcomas (both pediatric and adult), osteosarcomas.
4. Clinically significant gastrointestinal abnormalities which might interfere with oral dosing diagnosed as:

   * Active peptic ulcer disease.
   * Known intraluminal metastatic lesions with suspected bleeding.
   * Inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation.
   * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
   * Major resection of the stomach or small bowel.
5. Uncontrolled hypertension.
6. Unstable or serious concurrent condition (e.g., active infection requiring systemic therapy).
7. Prolongation of corrected QT interval (QTc) >480 msecs.
8. History of any one of more of the following cardiovascular conditions within the past 6 months:

   1. Cardiac angioplasty or stenting.
   2. Myocardial infarction.
   3. Unstable angina.
   4. Symptomatic peripheral vascular disease.
   5. Coronary artery by-pass graft surgery.
   6. Class II, III or IV congestive heart failure as defined by the New York Heart Association (NYHA).
   7. History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
9. Macroscopic hematuria
10. Haemoptysis that is clinically relevant within 4 weeks of first dose of study drug.
11. Evidence of active bleeding or bleeding diathesis.
12. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
13. Chemotherapy or radiation therapy within 2 weeks prior to the first dose of study drug.
14. Biological therapy or treatment with an investigational agent within 28 days or 5 half-lives, whichever is longer prior to the first dose of study drug.
15. Prohibited medications listed in the protocol for 14 days or five half-lives of a drug (whichever is longer) prior to Visit 1 and for the duration of the study should not be taken.
16. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib.
17. Pregnancy or lactating.
18. Hypothyroidism.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 14 weeks
  To study the safety and feasibility of adding 6 weeks of orally administered Pazopanib to 25 x 2Gy in 5 weeks preoperative radiotherapy in extremity or head and neck area soft tissue sarcoma patients (to identify the Dose Limiting Toxicity (DLT) and the Recommend Phase II Dose (RPTD) if pazopanib is added to 50 Gy pre-operatively)

SECONDARY OUTCOMES:
the exploration/feasibility of dynamic imaging | 14 weeks
  The secondary objective is to explore the feasibility to perform perfusion weighted MRI imaging regarding tumor respons to RT and neoangio genesis inhibitor by pazopanib.

CONTACTS AND LOCATIONS:
Overall Officials: Rick Haas, MD,PhD, Principal Investigator — NKI
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands